CLINICAL TRIAL: NCT03865199
Title: A Narrative Intervention to Decrease Individual Level Abortion Stigma: A Randomized Controlled Trial
Brief Title: A Narrative Intervention to Decrease Abortion Stigma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Planned Parenthood Federation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB18-1683
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Stigma, Social
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Intervention Model Description: Women aged 18 or older undergoing medical or surgical abortion at Planned Parenthood of Illinois will be eligible for inclusion in the study. Recruitment will occur two days a week, altering days of the week, and all patients seen on recruitment days not meeting exclusion criteria will be offered the opportunity to enroll after their confirmatory ultrasound. This will be a non-blinded 1:1 randomized controlled trial. Randomization will be done using a computer-generated randomization sequence. A research assistant will place study group assignment in a sealed, opaque, sequentially numbered envelope. This envelope will be opened by the researcher obtaining consent, who will not be involved in clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention arm will view a digital story on a tablet created by the research team, then respond to a writing prompt. A baseline abortion stigma and psychological distress survey will be taken at enrollment and then again at follow-up after 2-4 weeks.
  Interventions: Behavioral: Narrative Intervention
- Control Group (No Intervention): The control group will receive care as usual at the abortion clinic. A baseline abortion stigma and psychological distress survey will be taken at enrollment and then again at follow-up after 2-4 weeks.

INTERVENTIONS:
Behavioral: Narrative Intervention — Participants in the intervention group will first view a digital story on a tablet with headphones that will combine a fictional patient's abortion story with basic medical and social facts regarding abortion. After viewing the narrative, participants will be asked to write a narrative either on a tablet provided or on paper with the prompt: "Patients have different thoughts and feelings about their experiences when they have this procedure. Tell a story (about yourself or someone else, real or imaginary) that might help another patient feel supported."
  Arms: Intervention Group

SUMMARY:
Abortion stigma is pervasive in the United States. It operates across multiple levels, including the individual, community, and structural. While abortion itself does not cause mental health problems, due to stigma, women who undergo abortion are at risk of suffering negative psychological responses including thought suppression and isolation, which can result in psychological distress. Few intervention studies have addressed abortion stigma. Research in other disciplines, in particular mental health, has demonstrated the importance of self-validation in improved coping. Drawing from psychologists' use of writing in cognitive therapy and the discipline of Narrative Medicine's emphasis on narrative as a mechanism of healing, the proposed study attempts to test a novel intervention to reduce individual level abortion stigma. The study will be a randomized controlled trial evaluating a narrative intervention to reduce individual level abortion stigma. The principal research question is: can a narrative intervention that aims to positively frame the abortion experience decrease individual level abortion stigma? An additional research question is: will women who take part in a narrative intervention to reduce abortion stigma have improved psychological responses to the abortion? Women in the intervention group will view a digital story on a tablet intending to provide education and normalization and then respond to a writing prompt aimed at cognitive restructuring. The control group will receive care as usual.

DETAILED DESCRIPTION:
The proposed study will be a two-arm, non-blinded, 1:1 randomized controlled trial of a narrative intervention to reduce individual level abortion stigma that will be conducted at Planned Parenthood of Illinois (PPIL). The narrative intervention combines exposing patients to a digital narrative and then asking them to respond to a writing prompt, aiming first to normalize the abortion experience and then to help frame it in positive terms. Women randomized to the intervention will view a story created by the research team on a tablet using headphones. The story will be read by an actor and digitally recorded for playback by the participant. The narrative will combine a fictional patient's abortion story with basic medical and social facts regarding abortion. After viewing the narrative, the participant will be asked to write a narrative either on a tablet provided or on paper with the prompt: "Patients have different thoughts and feelings about their experiences when they have this procedure. Tell a story (about yourself or someone else, real or imaginary) that might help another patient feel supported." The goal behind this prompt is to allow the participant to write a narrative that is based in personal experience, but that provides the opportunity to mentally join a "virtual community" through the act of speaking to and helping another (theoretical) patient. Participants randomized to the intervention will complete the intervention during the visit, prior to meeting with an educator. Participants randomized to the control arm will receive regular care in the abortion clinic.

Stigma will be measured at baseline and 2-4 weeks following the intervention with the Individual Level Abortion Stigma Scale (ILAS), a scale that was developed to measure the impact of abortion stigma interventions. Four items from The Profile of Mood States- Short Form (POMS-SF) will be used to assess psychological distress at the abortion visit and again at follow-up. Pre- and post-intervention test scores between groups will be compared in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or older undergoing medical or surgical abortion at Planned Parenthood of Illinois (PPIL) will be eligible for inclusion. Inclusion criteria include having an intrauterine pregnancy, having a smart phone to be able to follow-up by text message 2-4 weeks after the clinic appointment, having no contraindications to an outpatient medication or surgical abortion that same day, and not meeting any exclusion criteria.

Exclusion Criteria:

* Exclusion criteria will include non-English speaking, no working telephone, and less than 5th grade education level.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Individual level abortion stigma | 4 weeks
  Difference in score on the Individual Level Abortion Stigma Scale (ILAS) between baseline and follow-up: The ILAS is a validated 20-item scale that measures individual level stigma with four subscales including: worries about judgment, isolation, self-judgment, and community condemnation. The ILAS has a maximum score of five; in the study that established validity of this scale, the mean score was 1.35 with a standard deviation of 0.63. A higher score indicates greater stigma and a lower score indicates lesser stigma, so a greater decrease in mean scores between baseline and follow-up seen in the intervention group as compared to the control group would indicate an effect of the narrative intervention.

SECONDARY OUTCOMES:
Psychological distress | 4 weeks
  Difference in score on a modified version of the Profile of Mood States- Short Form (POMS-SF) between baseline and follow-up: Given the length of the POMS-SF, only a few items will be tested. The shortened form is a 37-item questionnaire that asks subjects to rate various adjectives or mood states on a Likert Scale. In this study, the items used will be "sad," "discouraged," "confident," and "satisfied." The scale is scored by adding up the scores associated with negative responses and subtracting the scores associated with positive responses. The maximum score is 4, and the minimum score is zero. A lower score indicates a lower level of psychologic distress. While using only a few items of the POMS-SF has not been specifically validated, we believe that it will provide useful information to evaluate our secondary outcome of psychological distress without placing a significant time burden on participants.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD, Principal Investigator — University of Chicago
Locations (1):
- Planned Parenthood, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The data from this study will not be shared outside of the researchers involved in this protocol.

REFERENCES:
- [Result] Cockrill K, Upadhyay UD, Turan J, Greene Foster D. The stigma of having an abortion: development of a scale and characteristics of women experiencing abortion stigma. Perspect Sex Reprod Health. 2013 Jun;45(2):79-88. doi: 10.1363/4507913. Epub 2013 May 2. PMID 23750622
- [Result] Shacham S. A shortened version of the Profile of Mood States. J Pers Assess. 1983 Jun;47(3):305-6. doi: 10.1207/s15327752jpa4703_14. PMID 6886962